CLINICAL TRIAL: NCT02574871
Title: Data Collection for Identification of the Chronic Stress Presence in Healthy Adult Subjects
Brief Title: Data Collection for Stress Identification
Status: Completed | Type: Observational
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Annie France Frère Slaets, PhD, University of Mogi das Cruzes
Other Study IDs: 28201014.2.0000.5497
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Stress
Keywords: Stress; Chronic stress; Perceived stress; Psychological distress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single Group: Psychological and biological data collection
  Interventions: Other: Psychological and biological data collection

INTERVENTIONS:
Other: Psychological and biological data collection — Psychological and biological data collection for identification of the chronic stress presence

SUMMARY:
This study consists of psychological and biological data collection for identification of the chronic stress presence in healthy adult subjects. The psychological data collected were the results provided by three different instruments: ISSL, PSS and SRRS. The biological data collected were the blood pressure, the skin temperature, the galvanic skin response, and the heart rate variability in time and frequency domain.

DETAILED DESCRIPTION:
According to the WHO (World Health Organization) the stress has become a worldwide epidemic and has been considered as the disease of the century, attaining people of different ages and occupations. Stress is defined as a pressure or tension, of a physical, mental or emotional type, which overwhelms the individual and adversely affects the performance of his physical and intellectual functions. When stress is prolonged, the immune system is affected, leaving the body subject to disease and premature aging. Among the psychophysiological reactions associated with excessive stress are chronic fatigue, ulcers, depression, hypertension and heart attack. In light of these consequences, it is important that measures are taken to early identifying the symptoms of stress, allowing people to be properly treated and resume their normal activities.

The studies presented in literature suggest the possibility of using biological signals as indicators of the presence of stress. In these studies, certain physiological variables are measured and related to this stress on the individual. However, most previous studies focused on acute stress, meaning that short-lived. The objective of this study was to relate certain physiological indicators with the presence of chronic stress, ie that long-lasting and often not perceived by the individual.

To this end, the investigators performed the measurement of blood pressure values, skin temperature, galvanic skin response and heart rate variability, and compared with the results provided by the ISSL (Lipp's Inventory of Stress Symptoms for Adults), PSS (Perceived Stress Scale) and SRRS (Social Readjustment Rating Scale), as the stress condition of the individual. The heart rate variability was checked in both time and frequency domain. All of the physiological signals were monitored by non-invasive and non-intrusive sensors and totally safe for participants.

To investigate the relationship between the physiological variables and the existing chronic stress condition the investigators used an algorithm for analysis of biological signals based on Multilayer Perceptron Neural Network with Backpropagation Algorithm (MLP) and Principal Components Analysis (PCA). To evaluate the performance of the classifier on the identification of chronic stress the investigators check the indicators of precision, sensitivity, specificity and accuracy. The results were then analyzed by Receiver Operating Characteristic Curves (ROC).

Ethical approval was obtained from the Local Ethics Committee (CAAE-28201014.2.0000.5497) for the participants. They had been informed about the methodology and confidentiality of their personal information. All procedures were performed after written informed consent from all participants. Data collection was completed in October 2014.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Presence of any disease
* Use of medications to control blood pressure
* Use of anxiety medications and antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: undergraduate students
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 5 minutes
  Short-term heart rate variability recording, according to recommendations of the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology

SECONDARY OUTCOMES:
Blood pressure measurement (BP) | 1 minute
  Blood pressure measurement of volunteers, according to the guidelines of the Brazilian Society of Cardiology (SBC)
Temperature measurement (ST) | 5 minutes
  Skin temperature measurement of volunteers with a digital thermometer
Galvanic skin response (GSR) | 5 minutes
  Galvanic skin response of volunteers recording with a digital GSR recorder
Stress assessment (ISSL) | 10 minutes
  Stress assessment of volunteers, according to the Lipp's Inventory of Stress Symptoms for Adults (ISSL)
Perceived stress (PSS) | 5 minutes
  Perceived stress of volunteers, according to the Perceived Stress Scale (PSS)
Social stress (SRRS) | 5 minutes
  Social stress of volunteers, according to the Social Readjustment Rating Scale (SRRS)

CONTACTS AND LOCATIONS:
Overall Officials: Annie F Frere Slaets, PhD, Principal Investigator — University of Mogi das Cruzes

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Zhai J, Barreto A. Stress detection in computer users based on digital signal processing of noninvasive physiological variables. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:1355-8. doi: 10.1109/IEMBS.2006.259421. PMID 17946041
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Bandeira DR, Pawlowski J, Goncalves TR, Hilgert JB, Bozzetti MC, Hugo FN. Psychological distress in Brazilian caregivers of relatives with dementia. Aging Ment Health. 2007 Jan;11(1):14-9. doi: 10.1080/13607860600640814. PMID 17164153